CLINICAL TRIAL: NCT04685863
Title: Effect of Neurodynamic Mobilization Techniques on Knee Extension Range of Motion of Asymptomatic Young Students: a Prospective, Comparative Study.
Brief Title: Slump Physiotherapy : Effect on the physiologicAl Knee Extension Range-of-motion
Acronym: SPEAKER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/0251/OB
Record Dates: First submitted 2020-12-02; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Knee Extension
Keywords: Neurodynamic Mobilization Technique; Physiotherapy; SLUMP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mobilizing the knee with active neurodynamic sliding technique (active Slump slider) — 60 physiotherapy students perform measurements during three tutorials. The first involves training in evaluation techniques. The second involves mobilizing the knee, out of the SLUMP position. The third tutorial includes neuronal mobilization in SLUMP.
  Other Names: Mobilizing the knee, out of the SLUMP position

SUMMARY:
Background: The neurodynamics technique seems interesting for increased lower limb flexibility of the lower limbs in healthy subjects. The objective of this study is to assess the physiological effects of the SLUMP sliding technique on the range of knee extension during the SLUMP test.

Methods: 60 physiotherapy students perform measurements during three tutorials. The first involves training in evaluation techniques. The second involves mobilizing the knee, out of the SLUMP position. The third tutorial includes neuronal mobilization in SLUMP.

Knee extension in SLUMP position is measured immediately after completing techniques. The mobilization amplitudes (degrees) will be compared between the techniques by a Student test on paired series, each subject being his own control.

Discussion: The results of this study will provide evidence for the physiological effect of SLUMP sliding techniques performed by physiotherapy students on the range of knee extension during the SLUMP test in asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in second year of physiotherapy training in Rouen's physiotherapy Institute, taking part to neurodynamic technique course unit (CU 7)
* Ability to perform daily physiotherapy techniques, assessed by an accredited doctor from regional health agency and a medical examination during the first year of scholarship (occupational medicine service of Rouen's University hospital)
* French commonly spoken and red
* Aged 18 or older
* Registered to the national care & health system (Social security number)
* Willingness to take part to the study

Exclusion Criteria:

* Person denied of freedom by judicial or administrative decision
* Person requiring a guardian, guardianship or curators
* History of psychological disease/illness or sensorial disease preventing from understanding the recruitment conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are voluntary students, enrolled in second year of physiotherapy, taking part to a neurodynamic technique course unit (CU 7) in the Rouen Physiotherapy Institute. Data collection is performed during three practical works of CU 7.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2020-12-16 (Estimated); Study Completion 2020-12-16 (Estimated)

PRIMARY OUTCOMES:
Knee extension angle achieved in SLUMP test position: - after a control technique during the second practical work (TD2) | day 14 from inclusion
  degree
Knee extension angle achieved in SLUMP test position : - after neurodynamic sliding techniques in SLUMP during the third practical work (TD3) | day 21 from inclusion
  degree

SECONDARY OUTCOMES:
Finger-to-floor distance | days 14 and 21 from inclusion
  centimeter
Hamstring flexibility (passive knee extension test) | days 14 and 21 from inclusion
  degree
Angle of knee extension achieved in SLUMP test between "active neurodynamic technique" group and "passive neurodynamic technique" group | days 14 and 21 from inclusion
  degree

CONTACTS AND LOCATIONS:
Overall Officials: Timothée Gillot, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University hospital, Rouen, France